CLINICAL TRIAL: NCT00331760
Title: A Phase II Study of Intensity Modulated Radiation Therapy (IMRT) to the Pelvis ± Chemotherapy for Post-Operative Patients With Either Endometrial or Cervical Carcinoma
Brief Title: Intensity-Modulated Radiation Therapy to the Pelvis With or Without Chemotherapy in Treating Patients With Endometrial Cancer or Cervical Cancer That Has Been Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0418; CDR0000472905
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Cervical Cancer; Endometrial Cancer
Keywords: stage I endometrial carcinoma; stage II endometrial carcinoma; stage III endometrial carcinoma; endometrial adenoacanthoma; endometrial adenocarcinoma; endometrial adenosquamous cell carcinoma; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endometrial Cancer: IMRT (Other): Endometrial Cancer patients receive Intensity Modulated Radiation Therapy (IMRT) 28 fractions over 5.5 weeks.
  Interventions: Radiation: intensity-modulated radiation therapy
- Cervical Cancer: IMRT + Chemotherapy (cisplatin) (Other): Cervical patients receive Intensity Modulated Radiation Therapy (IMRT) 28 fractions over 5.5 weeks and concurrent weekly cisplatin 40 mg/m^2 for five weeks.
  Interventions: Drug: cisplatin; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: cisplatin
  Arms: Cervical Cancer: IMRT + Chemotherapy (cisplatin)
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Specialized radiation therapy (RT), such as intensity-modulated radiation therapy (IMRT), that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving intensity-modulated radiation therapy to the pelvis with or without chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well intensity-modulated radiation therapy to the pelvis with or without chemotherapy works in treating patients with endometrial cancer or cervical cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the transportability of intensity modulated radiotherapy (IMRT) to a multi-institutional setting in patients with resected endometrial or cervical cancer.
* Compare the efficacy, in terms of reducing short-term bowel injury, of IMRT versus standard treatments.
* Assess adverse events related to this regimen.
* Estimate the rates of local-regional control, distant metastasis, and disease-free and overall survival.
* Evaluate chemotherapy compliance with this regimen for patients with cervical carcinoma.

OUTLINE: This is a multicenter study. Patients are stratified according to diagnosis (cervical vs endometrial cancer).

All patients undergo intensity modulated radiotherapy (IMRT) once a day, 5 days a week, for 5.5 weeks. Patients with cervical cancer also receive cisplatin IV over 30-60 minutes on day 1 or 2. Treatment with cisplatin repeats every 7 days for 5 courses (during radiotherapy) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 6 weeks post-IMRT and then every 3 months for 2 years, every 6 months for years 3-5, and then annually for at least 3 years.

PROJECTED ACCRUAL: A total of 92 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must have undergone a hysterectomy (total abdominal, vaginal, radical, or laparoscopic-assisted vaginal) within 7 weeks prior to study entry

  * Patients with endometrial cancer must have also undergone a bilateral salpingo-oophorectomy
* Histologically confirmed diagnosis of 1 of the following:

  * Endometrial cancer meeting 1 of the following criteria:

    * Stage IB grade 3, IC grade 1-3, IIA, or IIB disease requiring postoperative pelvic radiotherapy
    * Unstaged (no lymph node dissection or sampling) stage IB grade 2 disease
    * Stage IIIC with all of the following:

      * Pelvic lymph node positive only
      * Para-aortic nodes sampled negative
      * Not receiving chemotherapy
  * Cervical cancer meeting 1 of the following criteria:

    * Post-radical hysterectomy and requires postoperative pelvic radiotherapy due to any of the following:

      * Positive pelvic nodes (negative para-aortic nodes)
      * Microscopic parametrial involvement and negative margins
      * Disease qualified by Sedlis criteria must have 2 of the following risk factors:

        * 1/3 or more stromal invasion
        * Lymph-vascular space invasion
        * Large clinical tumor diameter (≥ 4 cm)
    * Post-simple hysterectomy with negative margins and negative nodes by CT scan, MRI, or positron emission tomography-CT scan
* No requirement for extended-field radiotherapy beyond the pelvis
* No histologically confirmed papillary serous, clear cell, or neuroendocrine (either large or small cell) disease, endometrial stromal sarcoma, leiomyosarcoma, or malignant müllerian mixed tumor
* No evidence of metastatic disease outside of the pelvis
* No microscopic involvement of the resection margin (< 3 mm)

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* WBC (white blood cell count) ≥ 4,000/mm³ (cervical cancer patients only)
* Absolute neutrophil count ≥ 1,800/mm³ (cervical cancer patients only)
* Platelet count ≥ 100,000/mm³ (cervical cancer patients only)
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)
* Serum creatinine ≤ 2.0 mg/dL (cervical cancer patients only)
* Creatinine clearance ≥ 50 mL/min (cervical cancer patients only)
* AST (aspartate aminotransferase) ≤ 2 times upper limit of normal
* Bilirubin ≤ 2 times upper limit of normal
* Patients must not exceed the weight and size limits of the treatment table or CT scanner

  * No mental status changes or bladder control problems that would preclude study compliance with bladder-filling instructions
* No active inflammatory bowel disease
* No severe, active, concurrent illness, defined as any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring IV antibiotics
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * AIDS
* No history of allergy to cisplatin (cervical cancer patients)
* No prior invasive malignancy (except nonmelanoma skin cancer) unless disease-free for ≥ 3 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to the pelvis that would result in overlap of radiotherapy fields
* No prior platinum-based chemotherapy (cervical cancer patients)
* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], or pegfilgrastim)
* No concurrent prophylactic thrombopoietic agents
* No concurrent amifostine or other protective agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-03; Primary Completion 2009-02 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuja Jhingran, MD, Study Chair — M.D. Anderson Cancer Center
Locations (153):
- United States (151):
  - Auburn Radiation Oncology, Auburn, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Valley Medical Oncology, Fremont, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Bay Medical, Panama City, Florida
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Oncology Center at Saint Margaret Mercy Healthcare Center, Hammond, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Providence Medical Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Johnson County Radiation Therapy, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - South Suburban Oncology Center, Quincy, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - Kansas City Cancer Center at St. Joseph's Medical Mall, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Associates of Kansas City at Northland Radiation Oncology Center, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Radiation Oncology Associates, PA, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Cancer Institute of New Mexico, Santa Fe, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Huron Hospital Cancer Care Center, Cleveland, Ohio
  - Euclid Hospital, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital Cancer Care Center, Warrensville Heights, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec

REFERENCES:
- [Result] Jhingran A, Winter K, Portelance L, Miller B, Salehpour M, Gaur R, Souhami L, Small W Jr, Berk L, Gaffney D. A phase II study of intensity modulated radiation therapy to the pelvis for postoperative patients with endometrial carcinoma: radiation therapy oncology group trial 0418. Int J Radiat Oncol Biol Phys. 2012 Sep 1;84(1):e23-8. doi: 10.1016/j.ijrobp.2012.02.044. Epub 2012 Apr 28. PMID 22543211

RESULTS

PARTICIPANT FLOW:
Groups:
- Endometrial Cancer: IMRT: Endometrial Cancer patients receive Intensity Modulated Radiation Therapy (IMRT)
- Cervical Cancer: IMRT + Chemotherapy (Cisplatin): Cervical patients receive Intensity Modulated Radiation Therapy (IMRT) + Chemotherapy (cisplatin)
Period: Overall Study
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Started | 58 | 48
Completed | 43 (Subjects contributing data to the primary analysis are considered to have completed the study.) | 40
Not Completed | 15 | 8
Not completed — Ineligible / no protocol treatment | 15 | 8

BASELINE CHARACTERISTICS:
Population: All registered patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin) | Total
Number analyzed (Participants) | 58 | 48 | 106
Age, Continuous [Median (Full Range); unit: years] | 58 [36 to 84] | 43 [22 to 71] | 53 [22 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 48 | 106
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Reproducibility of Radiation Technique (Number of Unacceptable Deviations in Central IMRT Quality Assurance Review)
Description: Central quality assurance review of the IMRT planning and dosing categorized unacceptable deviations (UD) from protocol compliance with the delineation of planning target volume for the vagina and pelvic lymph nodes. Each arm of this study is considered independently, they are not compared to each other. The study was designed such that, for each arm, 5 or more of 42 subjects scored as unacceptable would determine the respective treatment technique as not reproducible. For each arm this design provides 90% power with a 0.05 type I error to reject the null hypothesis that the true probability of concluding the given technique to be reproducible is <= 80%. The alternative hypothesis is that the true probability is >= 95%.
  For [vagina / pelvic lymph nodes]: UD is defined as: The 90% isodose surface covers < 95% of [internal target volume (ITV)/ planned target volume (PTV)] 50.4 or > 5% of the [ITV/PTV] 50.4 receives over 115%.
Time Frame: IMRT planning and dosing data is centrally reviewed for quality assurance after treatment delivery.
Population: All eligible patients.
Measure: Number; unit: participants
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Number analyzed (Participants) | 43 | 40
participants | 1 | 0

2. Secondary Outcome: Percentage of Patients With Grade 2+ Bowel Adverse Events
Description: Bowel adverse events are defined as any of the following adverse events: diarrhea; enteritis; fistula; ileus:gastrointestinal (GI); incontinence:anal; necrosis:GI; obstruction:GI; perforation:GI; proctitis; stricture/stenosis (including anastomotic):GI. Adverse events are graded using Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the adverse event (AE). The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to adverse event.
Time Frame: From the start of treatment to 90 days.
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Number analyzed (Participants) | 43 | 40
percentage of participants | 27.9 [16.6 to 42.8] | 22.5 [12.1 to 37.7]
Statistical Analysis 1: Comparison: Endometrial Cancer: IMRT; A sample size of 42 patients provides 64% power to detect a reduction in short-term grade 2 or higher bowel AEs from historical rate of 40% to 25%; Test type: Superiority; p = 0.12, Chi-squared
Statistical Analysis 2: Comparison: Cervical Cancer: IMRT + Chemotherapy (Cisplatin); A sample size of 42 patients provides 88% power to detect a reduction in short-term grade 2 or higher bowel AEs from historical rate of 40% to 20%; Test type: Superiority; p = 0.043, Chi-squared

3. Secondary Outcome: Percentage of Patients With Any Grade 3+ Treatment-related Adverse Events
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the adverse event (AE). The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE.
Time Frame: From start of treatment to the end of follow-up. Maximum follow-up at time of analysis was 10.2 years for endometrium cancer patients and 9.5 years for cervical cancer patients.
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Number analyzed (Participants) | 43 | 40
percentage of participants
  Non-hematologic | 19 [9 to 33] | 30 [18 to 46]
  Overall | 30 [19 to 45] | 48 [33 to 63]

4. Secondary Outcome: Percentage of Patients With Any Late Grade 3+ Treatment-related Adverse Events
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each adverse events (AE) based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE. Late is defined as more than 90 days after the start of radiation therapy.
Time Frame: From 91 days after start of study treatment to the end of follow-up. Maximum follow-up at time of analysis was 10.2 years for endometrium cancer patients and 9.5 years for cervical cancer patients.
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Number analyzed (Participants) | 43 | 40
percentage of participants
  Non-hematologic | 12 [5 to 25] | 10 [3 to 24]
  Overall | 12 [5 to 25] | 10 [3 to 24]

5. Secondary Outcome: Percentage of Cervical Carcinoma Patients That Were Chemotherapy Compliant
Description: Chemotherapy treatment was centrally reviewed for quality assurance and compliance once complete chemotherapy treatment data was received from sites.
Time Frame: From start to end of chemotherapy, approximately five weeks from registration.
Population: Eligible patients in the chemotherapy group (cervical cancer patients) who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Number analyzed (Participants) | 40
percentage of participants | 80 [65 to 90]

6. Secondary Outcome: Rate of Local-regional Failure at Five Years
Description: Local-regional failure time is defined as time from registration to date of local-regional failure (any failure in the treatment field, which will be the pelvis only), death without local-regional failure (competing risk), or last known follow-up (censored). Local-regional failure rates are estimated by the cumulative incidence method.
Time Frame: From registration to five years.
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Number analyzed (Participants) | 43 | 40
percentage of participants | 5 [1 to 14] | 8 [2 to 19]

7. Secondary Outcome: Rate of Distant Metastases at Five Years
Description: Distant Metastases failure time is defined as time from registration to date of distant disease, death without distant metastases (competing risk), or last known follow-up (censored) and is estimated by the cumulative incidence method. Para-aortic nodal disease is considered to be distant disease for a cervical primary, but not for an endometrial primary.
Time Frame: From registration to five years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Number analyzed (Participants) | 43 | 40
percentage of participants | 7 [2 to 17] | 14 [5 to 27]

8. Secondary Outcome: Rate of Disease-free Survival at Five Years
Description: Disease-free survival time is defined as time from registration to date of failure (any tumor recurrence, development of distant metastases or death from any cause) and is estimated by the Kaplan-Meier method. Patients last known to be alive without failure are censored at the date of last contact.
Time Frame: From registration five years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Number analyzed (Participants) | 43 | 40
percentage of participants | 88 [74 to 95] | 84 [68 to 92]

9. Secondary Outcome: Rate of Overall Survival at Five Years
Description: Overall survival time is defined as time from randomization to the date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From randomization to five years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Number analyzed (Participants) | 43 | 40
percentage of participants | 88 [74 to 95] | 92 [77 to 97]

ADVERSE EVENTS:
Description: Eligible patients who started study treatment are included. Patients experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Endometrial Cancer: IMRT | Cervical Cancer: IMRT + Chemotherapy (Cisplatin)
Serious Adverse Events (participants affected / at risk) | 2/43 | 3/40
Other Adverse Events (participants affected / at risk) | 42/43 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endometrial Cancer: IMRT (N=43) | Cervical Cancer: IMRT + Chemotherapy (Cisplatin) (N=40)
Diarrhoea NOS (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Urinary tract infection NOS (Infections and infestations) | 1 | 0
Lymphopenia (Investigations) | 0 | 1
Neutrophil count (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Endometrial Cancer: IMRT (N=43) | Cervical Cancer: IMRT + Chemotherapy (Cisplatin) (N=40)
Hemoglobin (Blood and lymphatic system disorders) | 11 | 21
Hearing impaired (Ear and labyrinth disorders) | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 5
Abdominal distention (Gastrointestinal disorders) | 1 | 3
Abdominal pain NOS (Gastrointestinal disorders) | 12 | 10
Anal discomfort (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 5 | 8
Diarrhoea NOS (Gastrointestinal disorders) | 33 | 33
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 6 | 2
Flatulence (Gastrointestinal disorders) | 1 | 2
Gastritis NOS (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 14 | 27
Proctitis NOS (Gastrointestinal disorders) | 1 | 5
Vomiting NOS (Gastrointestinal disorders) | 1 | 14
Fatigue (General disorders) | 20 | 27
Pain NOS (General disorders) | 3 | 1
Gingival infection (Infections and infestations) | 0 | 2
Urinary tract infection NOS (Infections and infestations) | 0 | 3
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 6 | 6
Fracture NOS (Injury, poisoning and procedural complications) | 2 | 2
Radiation recall syndrome (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 4 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 2
Blood bilirubin increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 0 | 3
Leukopenia NOS (Investigations) | 17 | 26
Lymphopenia (Investigations) | 9 | 18
Neutrophil count (Investigations) | 3 | 5
Platelet count decreased (Investigations) | 7 | 11
Weight decreased (Investigations) | 4 | 5
Anorexia (Metabolism and nutrition disorders) | 4 | 9
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 10 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 5
Hypokalemia (Metabolism and nutrition disorders) | 5 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 6
Hyponatremia (Metabolism and nutrition disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 6
Headache (Nervous system disorders) | 0 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 5
Agitation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 6
Depression (Psychiatric disorders) | 7 | 3
Insomnia (Psychiatric disorders) | 0 | 6
Libido decreased (Psychiatric disorders) | 3 | 3
Bladder spasm (Renal and urinary disorders) | 0 | 3
Cystitis NOS (Renal and urinary disorders) | 3 | 7
Pollakiuria (Renal and urinary disorders) | 10 | 10
Urethral pain (Renal and urinary disorders) | 1 | 3
Urinary incontinence (Renal and urinary disorders) | 9 | 7
Urinary retention (Renal and urinary disorders) | 1 | 4
Pelvic pain NOS (Reproductive system and breast disorders) | 3 | 5
Vaginal atresia (Reproductive system and breast disorders) | 6 | 14
Vaginal discharge (Reproductive system and breast disorders) | 3 | 8
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 4
Vaginal pain (Reproductive system and breast disorders) | 2 | 4
Vaginal stricture (Reproductive system and breast disorders) | 3 | 0
Vaginitis (Reproductive system and breast disorders) | 3 | 2
Vulvovaginal dryness (Reproductive system and breast disorders) | 4 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 2
Telangiectasia (Skin and subcutaneous tissue disorders) | 3 | 2
Hot flushes NOS (Vascular disorders) | 4 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No